CLINICAL TRIAL: NCT06263218
Title: Single-center, Non-interventional, Retrospective Study on the Outcomes of Infection by CMV, Treatment Patterns, and Healthcare Resource Utilization Among CMV Recipients Kidney Transplant in Brazil
Brief Title: Real-world CMV Outcomes Among Kidney Transplant Recipients in Brazil
Status: Enrolling by invitation | Type: Observational
Sponsor: Hospital do Rim e Hipertensão (Other)
Responsible Party: Principal Investigator, Helio Tedesco Silva Junior, Principal investigator, Hospital do Rim e Hipertensão
Other Study IDs: CCR-2023-200344
Record Dates: First submitted 2023-09-21; First posted 2024-02-16 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: CMV Infection; CMV Viremia
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a single-center, non-interventional, retrospective study of data, at the level of the individual without identification, extracted from medical records of adult patients undergoing a kidney transplant procedure after 1st from January 2018 until reaching the sample size enrollment (around 500 individuals); this refers to the period of verification of individuals' eligibility for entry into the study. Individuals under strategy preemptive patients who developed CMV infection/disease within 12 months after transplantation. The data will be collected from date of transplant (including pre-transplant clinical history) until completion of at least 12 months after transplantation, or until graft loss, or recipient death or loss to follow-up, when/if applicable.

DETAILED DESCRIPTION:
Data will be collected from medical records and will include transplant recipient characteristics, transplant-related information, CMV status, clinical outcomes, treatment patterns, healthcare resource utilization and captured on an electronic Intake Form.

Study-specific Case Report (eCRF) The sponsor will create a Statistical Analysis Plan (SAP) before collection begins of data. The eCRF system will comply with research regulations

ELIGIBILITY:
Inclusion Criteria:

* Received a single kidney transplant after January 1, 2018
* Age over 18 years at time of kidney transplant.
* It was under preemptive strategy.
* Diagnosed with CMV infection/disease within the first 12 months after kidney transplant.
* Follow-up information is available in medical records for at least 12 months after confirmation of CMV infection, or even loss of the allograft, death of the recipient or loss of follow-up of the receiver, when/if applicable.

Exclusion Criteria:

* Diagnosed as a carrier of the human immunodeficiency virus (HIV+), hepatitis B virus and/or hepatitis C before kidney transplantation.
* Participation in any interventional study during the period between kidney transplantation and a period of 12 months after CMV diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be entirely adult kidney transplant recipients (age ≥18 years at the time of time of transplantation) who developed a first episode of CMV infection/disease in the first year of transplant. Eligible individuals will be enrolled consecutively based on transplant date, starting from the first year as defined in the inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-12-29 (Estimated)

PRIMARY OUTCOMES:
Incidence of infection, CMV disease, and tissue invasive disease. | 12 months
  Incidence of infection, CMV disease, and tissue invasive disease.

SECONDARY OUTCOMES:
Incidence recurrent CMV infection/disease | 12 months
  Incidence recurrent CMV infection/disease
Incidence of refractory CMV infection/disease | 12 months
  Incidence of refractory CMV infection/disease

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital do Rim, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No